CLINICAL TRIAL: NCT04201431
Title: A Phase I/IIa Clinical Trial to Assess the Safety, Immunogenicity and Efficacy of the Blood-stage Plasmodium Vivax Malaria Vaccine Candidate PvDBPII in Matrix M1 in Healthy Adults Living in the UK
Brief Title: Safety, Immunogenicity and Efficacy of the Blood-stage Plasmodium Vivax Malaria Vaccine Candidate PvDBPII in Matrix M1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: VAC079
Record Dates: First submitted 2019-11-18; First posted 2019-12-17 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2022-09

CONDITIONS: Malaria, Vivax
Keywords: PvDBPII
MeSH Terms: conditions — Malaria, Vivax | interventions — Matrix-M

STUDY DESIGN:
Intervention Model Description: Group 2 is optional to be added only if fewer than 8 volunteers complete in Group 1.
  Up to 6 volunteers from Group 1 will be invited to join Group 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Up to 12 volunteers in Group 1 will receive three doses of the PvDBPII 50ug/Matrix M1 50ug candidate vaccine at 1, 2 and 12-18 months prior to blood-stage CHMI 2-4 weeks after the third vaccination.
  Interventions: Biological: PvDBPII/Matrix-M1
- Group 2 (Experimental): If fewer than 8 volunteers complete the study in Group 1, then new volunteers will be recruited into Group 2, to make up a total of 10 to 12 volunteers who complete 3 vaccinations and CHMI between Groups 1 and 2. Group 2 volunteers will receive three doses of the PvDBPII 50ug/Matrix M1 50ug candidate vaccine at monthly intervals, prior to blood-stage CHMI 2-4 weeks after the third vaccination.
  Interventions: Biological: PvDBPII/Matrix-M1
- Group 3 (Experimental): Up to 6 volunteers from Group 1 will receive a fourth dose of PvDBPII 50ug/Matrix M1 50ug, at 5 months post the third dose, prior to a second CHMI 2-4 weeks later.
  Interventions: Biological: PvDBPII/Matrix-M1

INTERVENTIONS:
Biological: PvDBPII/Matrix-M1 — 50ug PvDBPII in 50ug Matrix M1

SUMMARY:
This is an Open label, first-in-human, Phase I/IIa, blood-stage P. vivax malaria vaccine trial to assess the safety, immunogenicity and efficacy of the blood-stage Plasmodium vivax malaria vaccine candidate PvDBPII in Matrix M1 in healthy adults living in the UK.

DETAILED DESCRIPTION:
This Phase I/IIa clinical trial is designed to primarily assess the safety of the PvDBPII-Matrix M1 vaccine in healthy volunteers and to establish whether the PvDBPII-Matrix M1 vaccine can demonstrate a reduced parasite multiplication rate in vaccinated subjects compared to infectivity controls in a blood-stage controlled human malaria infection model.

Up to 24 healthy volunteers aged 18-45 will be recruited in England at the Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Oxford.

Volunteers in Groups 1 and 2 will receive three doses of the PvDBPII 50ug/Matrix M1 50ug candidate vaccine prior to blood-stage CHMI 2-4 weeks after the third vaccination. Volunteers in Group 1 who complete 3 vaccinations and CHMI will be invited back for a fourth vaccination at 5 months following their third vaccination and form a new study group- Group 3.

Volunteers will undergo blood stage CHMI with Plasmodium vivax.

Volunteers in a parallel study (VAC069), who will undergo the same CHMI without prior vaccination, will be used as infectivity controls.

Participants in Group 1 will be followed for approximately 9 months after the third vaccination, approximately 2 years in total from enrolment. Participants in Group 2 will be followed for 1 year from enrolment. Participants in Group 3 will be followed for 9 months after their final (fourth) vaccination, approximately up to 2.5 years in total from enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 45 years.
* Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
* Normal serum levels of Glucose-6-phosphate dehydrogenase (G6PD).
* Negative haemoglobinopathy screen
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Willing to allow the Investigators to discuss the volunteer's medical history with their General Practitioner.
* Women only: Must practice continuous highly effective contraception* for the duration of the study
* Agreement to permanently refrain from blood donation
* Written informed consent to participate in the trial.
* Reachable (24/7) by mobile phone during the period between CHMI and completion of all antimalarial treatment.
* Willing to take a curative anti-malarial regimen following CHMI.
* Willing to reside in Oxford for the post-challenge period, until antimalarials have been completed.
* Answer all questions on the informed consent quiz correctly at first or second attempt

  * Female volunteers are required to use a highly effective form of contraception during the course of the study as malaria challenge could pose a serious risk to both maternal health and the unborn foetus.

Exclusion Criteria:

* History of clinical malaria (any species).
* Travel to a clearly malaria endemic locality during the study period or within the preceding six months.
* Use of systemic antibiotics with known antimalarial activity within 30 days of CHMI (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* Use of anti-malarials within 30 days of CHMI
* Weight less than 50kg, as measured at the screening visit
* Receipt of immunoglobulins within the three months prior to planned administration of the vaccine candidate.
* Receipt of blood products (e.g., blood transfusion) at any time in the past.
* Peripheral venous access unlikely to allow twice daily blood testing (as determined by the Investigator).
* Receipt of an investigational product in the 30 days preceding enrolment, or planned receipt during the study period.
* Receipt of any vaccine in the 30 days preceding enrolment, or planned receipt of any other vaccine within 30 days preceding or following each study vaccination, with the exception of licensed COVID-19 vaccines, which should not be received between 14 days before to 7 days after any study vaccination
* Planned receipt of a COVID-19 vaccine between 2 weeks before the day of CHMI until completion of antimalarial treatment
* Concurrent involvement in another clinical trial or planned involvement during the study period
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine e.g. egg products, Kathon
* History of allergic disease or reactions likely to be exacerbated by malaria infection.
* History of clinically significant contact dermatitis
* Any history of anaphylaxis in reaction to vaccinations
* Pregnancy, lactation or intention to become pregnant during the study.
* Use of medications known to cause prolongation of the QT interval and existing contraindication to the use of Malarone.
* Use of medications known to have a potentially clinically significant interaction with Riamet and Malarone.
* Any clinical condition known to prolong the QT interval.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Disturbances of electrolyte balance, e.g. hypokalaemia or hypomagnesaemia.
* Family history of congenital QT prolongation or sudden death.
* Contraindications to the use of both of the proposed anti-malarial medications; Riamet Malarone.
* History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ).
* History of serious psychiatric condition that may affect participation in the study.
* Any other serious chronic illness requiring hospital specialist supervision.
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 25 standard UK units every week.
* Suspected or known injecting drug abuse in the 5 years preceding enrolment.
* Hepatitis B surface antigen (HBsAg) detected in serum.
* Seropositive for hepatitis C virus (antibodies to HCV) at screening or (unless has taken part in a prior hepatitis C vaccine study with confirmed negative HCV antibodies prior to participation in that study, and negative HCV RNA PCR at screening for this study).
* Positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
* Volunteers unable to be closely followed for social, geographic or psychological reasons.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urinalysis or clinical examination. In the event of abnormal test results, confirmatory repeat tests will be requested. Procedures for identifying laboratory values meeting exclusion criteria are shown in SOP VC027.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data.
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Exclusion criteria on day of CHMI

The following constitute absolute contraindications to CHMI:

* Acute disease, defined as moderate or severe illness with or without fever
* Current COVID-19 infection, defined as ongoing symptoms with positive COVID-19 PCR swab test taken during current illness or positive COVID-19 PCR swab test within preceding 14 days without symptoms.
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Minassian, Dr, Principal Investigator — Jenner Institute
Locations (1):
- CCVTM, University of Oxford, Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou MM, Barrett JR, Themistocleous Y, Rawlinson TA, Diouf A, Martinez FJ, Nielsen CM, Lias AM, King LDW, Edwards NJ, Greenwood NM, Kingham L, Poulton ID, Khozoee B, Goh C, Mac Lochlainn DJ, Salkeld J, Guilotte-Blisnick M, Huon C, Mohring F, Reimer JM, Chauhan VS, Mukherjee P, Biswas S, Taylor IJ, Lawrie AM, Cho JS, Nugent FL, Long CA, Moon RW, Miura K, Silk SE, Chitnis CE, Minassian AM, Draper SJ. Impact of a blood-stage vaccine on Plasmodium vivax malaria. medRxiv [Preprint]. 2022 May 30:2022.05.27.22275375. doi: 10.1101/2022.05.27.22275375. PMID 35664997

RESULTS

PARTICIPANT FLOW:
Period: Vaccinations and Primary CHMI
Arm/Group | Group 1 | Group 2 | Group 3
Started | 12 | 4 | 0
Completed | 6 | 4 | 0
Not Completed | 6 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0
Period: 4th Vaccination and Secondary CHMI
Arm/Group | Group 1 | Group 2 | Group 3
Started | 0 | 0 | 5
Completed | 0 | 0 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group 3 participants are a subset 5 participants from Group 1 who completed 3 vaccinations and primary CHMI and subsequently received a 4th vaccination and secondary CHMI. Group 3 participants are therefore not separately shown here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 12 | 4 | 16
Age, Continuous [Mean (Full Range); unit: years] | 30 [19 to 44] | 35 [27 to 39] | 30 [19 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 2 | 12
  Male | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 11 | 4 | 15
  Ethnicity: Mixed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of the PvDBPII-Matrix M1 Vaccine Candidate, Assessed Through Collection of Data on the Frequency, Duration and Severity of Solicited and Unsolicited Adverse Events.
Description: Number of volunteers reporting a grade 3 solicited or unsolicited adverse event within 28 days post-vaccination or serious adverse event throughout the study period
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 12 | 4 | 5
Participants | 0 | 0 | 0

2. Primary Outcome: Establish Whether the PvDBPII-Matrix M1 Vaccine Can Demonstrate a Reduced Parasite Multiplication Rate in Vaccinated Subjects Compared to Infectivity Controls in a Blood-stage Controlled Human Malaria Infection Model
Description: Assessed by quantitative PCR-derived parasite multiplication rate (PMR). The PMR of the volunteers vaccinated with PvDBPII-Matrix M1 will be compared to the PMR of the malaria-naïve controls partaking in parallel primary CHMI in study VAC069.
Time Frame: 12 months
Population: Number of participants analyzed corresponds to participants undergoing primary CHMI. (Group 3 participants underwent secondary CHMI and therefore not included in this analysis.)
Measure: Median (Full Range); unit: parasite multiplication rate per 48hr
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 6 | 4
parasite multiplication rate per 48hr | 3.2 [2.3 to 4.3] | 6.3 [5.1 to 7.9]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Comparison of parasite multiplication rate in vaccinated subjects compared to infectivity controls in a blood-stage controlled human malaria infection model; Test type: Other — Comparison of pooled data from Groups 1 and 2 volunteers who completed primary CHMI with pooled data of infectivity controls undergoing primary CHMI from VAC069 study running in parallel (NCT03797989); p = 0.01, Wilcoxon (Mann-Whitney) — Two tailed p value reported for Mann-Whitney test comparing infectivity controls with vaccinees

3. Secondary Outcome: Assessment of the Humoral Immunogenicity of the PvDBPII-Matrix M1 Vaccine Candidate.
Description: Total IgG antibody response to the P. vivax Duffy-binding protein (PvDBPII) vaccine
Time Frame: 12 months
Population: Peak antibody response at 14 days after the third vaccination in volunteers who received three doses in Group 1 compared to Group 2. Group 3 participants were a subset of 5 participants from Group 1 who went on to complete a fourth vaccination and timepoints after the fourth vaccination are not directly comparable to timepoints after the third vaccination in Group 1 and Group 2 participants.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 4
μg/mL | 197.6 [153.1 to 335.3] | 52.64 [20.99 to 101.5]

4. Secondary Outcome: Assessment of the Cellular Immunogenicity of the PvDBPII-Matrix M1 Vaccine Candidate.
Description: PvDBPII-specific CD4+ CD45RA- CCR7- effector memory T cells producing IFN-γ at 14 days after the third vaccination
Time Frame: 12 months
Population: Peak T cell response at 14 days after the third vaccination in volunteers who received three doses in Group 1 and Group 2. Group 3 participants were a subset of 5 participants from Group 1 who went on to complete a fourth vaccination and timepoints after the fourth vaccination are not directly comparable to timepoints after the third vaccination in Group 1 and Group 2 participants.
Measure: Mean (Full Range); unit: percentage of IFN-γ+ cells
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 8 | 4
percentage of IFN-γ+ cells | 0.2951 [0.05600 to 0.9140] | 0.04350 [0.01400 to 0.05800]

5. Secondary Outcome: Immunological Readouts for Association With a Reduced Parasite Multiplication Rate
Description: Correlation between anti-PvDBP responses induced by the PvDBPII-Matrix M1 vaccine candidate and PMR.
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Assess the Durability of Any Reduction in PMR in Group 3 Volunteers Undergoing a Fourth Vaccination and Rechallenge
Description: Assessed by quantitative PCR-derived parasite multiplication rate (PMR). Comparison will be made between volunteers in Group 3 and two control groups: malaria-naive controls undergoing primary CHMI and volunteers undergoing their second CHMI in the parallel VAC069 study (NCT03797989).
Time Frame: 12 months
Measure: Median (Full Range); unit: parasite multiplication rate per 48hr
Arm/Group | Group 3
Number analyzed (Participants) | 5
parasite multiplication rate per 48hr | 4.3 [3.7 to 5.5]

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited adverse events were collected for 28 days following each vaccination. Serious adverse events were collected throughout the study duration: up to 29 months for Group 1, 12 months for Group 2 and 30 months for Group 3.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 8/12 | 3/4 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=12) | Group 2 (N=4) | Group 3 (N=5)
headache (Nervous system disorders) | 5 | 2 | 0
fatigue (General disorders) | 3 | 2 | 1
backpain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/31/NCT04201431/Prot_000.pdf